CLINICAL TRIAL: NCT02996539
Title: Heart Rate Variability and Diabetic Kidney Disease in Type 2 Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: Shi wei, MM (Other)
Responsible Party: Sponsor-Investigator, Shi wei, MM, Director, First People's Hospital of Kunming
Organization: First People's Hospital of Kunming (Other)
Other Study IDs: FirstPHKunming
Record Dates: First submitted 2016-11-24; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Type 2 diabetes: With Clinical examination and laboratory measurements
  Interventions: Other: Clinical examination and laboratory measurements

INTERVENTIONS:
Other: Clinical examination and laboratory measurements — Subjects were interviewed by a physician regarding their medical history, history of hypoglycemic attacks, smoking status, and alcohol consumption. Concentrations of blood urea nitrogen (BUN) and serum creatinine (SCr) were analyzed by the urease-ultraviolet rate method and picric acid method, respectively. Serum uric acid was determined using the enzymatic colorimetric method. Serum hemoglobin A1c (HbA1c) was measured by liquid enzymatic assay. Urine albumin and urine creatinine were found through immune turbidimetric analysis and the enzymatic method, respectively.
  Other Names: Physical examination and blood urine samples collection

SUMMARY:
Several studies have investigated an association between cardiac autonomic neuropathy (CAN) and albuminuria, glomerular filtration rate, or both, and hypothesized that CAN is involved in the pathogenesis of nephropathy. However, most of these studies had focused on Caucasians and were limited to a small number of patients with type 1 diabetes mellitus, or had used a conventional Ewing battery of tests based on dynamic cardiovascular maneuvers.Yet, there is consistent data showing that Asian diabetic populations, including the Chinese, have a higher risk of renal complications than Caucasians do.

The present study investigated an association between heart rate variability (HRV) parameters and diabetic kidney disease (DKD) in Chinese type 2 diabetes mellitus (T2DM) patients, specifically through time and frequency domain analyses of HRV and urine albumin creatinine ratio (UACR) or estimated glomerular filtration rate (eGFR).

DETAILED DESCRIPTION:
present study investigated an association between HRV parameters and DKD in Chinese T2DM patients, specifically through time and frequency domain analyses of HRV and UACR or eGFR

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM
* Adult patients has had consecutively undergone 24-hour Holter monitoring for heart rate variability analysis

Exclusion Criteria:

* Patients with acute complications of DM including diabetic ketoacidosis, hyperosmolar coma
* Foot ulcer
* Severe acute or chronic infection
* Chronic liver disease
* Dialysis or renal transplantation
* The presence of any serious concomitant disease affecting life expectancy were not eligible for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 392 patients of T2DM consecutively recruited from February 2013 to April 2015 in the inpatient department of Kunming First People's Hospital.The Institutional Review Board of Kunming First People's Hospital approved the study protocol. Adult patients with T2DM who had consecutively undergone 24-hour Holter monitoring for HRV analysis were included.
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Association between HRV and renal function (eGFR and UACR) | 1week
  Assessment of HRV HRV measurement based on 24-hour ambulatory ECG monitoring was obtained from all patients using a 3- channel digital Holter recorder (CB-2302-A, Wuxi, Jiangsu, China). Assessment of DKD DKD was defined as the presence of albuminuria (UACR ≥ 30 mg/g,urine albumin in milligram,creatinine in gram) or eGFR < 60 mL/min/1.73 m^2 (creatinine concentration in umol/l,creatinine molecular weight in micromole, volume in litre;urine volume per minute in milliliter per minute; body surface area in square meter) based on SCr levels. Albuminuria was defined using UACR of a single early-morning urine measurement.For all Participants, 132 patients had albuminuria and 50 patients with eGFR < 60 mL/min/1.73 m^2

SECONDARY OUTCOMES:
Clinical characteristics of patients | 1week
  Clinical examination and laboratory measurements Subjects were interviewed by a physician regarding their medical history, history of hypoglycemic attacks, smoking status, and alcohol consumption. A trained examiner measured the height (in meters) and body weight (in kilograms) of the patients. Body mass index (BMI) in kg/m^2, weight in kilograms, height in meters. Hypertension was defined as systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg, or both, or if the patient was already taking anti-hypertensive drugs. Blood and urine samples were analyzed at the medical examination center of Kunming First People's Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolei Chen, MM, Study Chair — Kunming first people's hospital
Locations (1):
- Internal medicine department, Kunming First People's Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes
The basic records of patients

REFERENCES:
- [Background] Tuttle KR, Bakris GL, Bilous RW, Chiang JL, de Boer IH, Goldstein-Fuchs J, Hirsch IB, Kalantar-Zadeh K, Narva AS, Navaneethan SD, Neumiller JJ, Patel UD, Ratner RE, Whaley-Connell AT, Molitch ME. Diabetic kidney disease: a report from an ADA Consensus Conference. Diabetes Care. 2014 Oct;37(10):2864-83. doi: 10.2337/dc14-1296. PMID 25249672
- See also: test link — http://www.cma.org